CLINICAL TRIAL: NCT03488810
Title: Radiotherapy and 6-month Androgen Deprivation Therapy With or Without Apalutamide in Intermediate and Limited High Risk Localized Prostate Cancer: a Phase III Study
Brief Title: Apalutamide With Radiotherapy and Androgen Deprivation Therapy in Prostate Cancer
Acronym: ARN-509
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Extended study timelines and additional budget could no longer be supported.
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1531-ROG
Record Dates: First submitted 2018-03-27; First posted 2018-04-05 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Apalutamide Prostate Cancer Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; apalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: ADT + radiation therapy (Active Comparator): Patient will receive 2 injections of a three-monthly LHRH agonist depot plus non-steroidal anti-androgen (rescue treatment) (e. g. flutamide, bicalutamide) PO daily for 4 weeks, started 2 weeks before the first LHRH agonist injection.
  All patients will receive standard fractionation radiation therapy (RT) between 0 and 12 weeks after first injection of LHRH agonist.
  Interventions: Other: Radiation Therapy; Drug: Luteinising Hormone Releasing Hormone analog agonist (LHRHa); Drug: Non-steroidal anti-androgen
- Arm B: ADT + radiation therapy + Apalutamide (Experimental): Patients will receive 2 injections of a three-monthly LHRH agonist depot. Apalutamide treatment: 240 mg PO daily, started the same day as the first LHRHa injection, for 6 months.
  All patients will receive standard fractionation radiation therapy (RT) between 0 and 12 weeks after first injection of LHRH agonist.
  Interventions: Other: Radiation Therapy; Drug: Apalutamide; Drug: Luteinising Hormone Releasing Hormone analog agonist (LHRHa)

INTERVENTIONS:
Other: Radiation Therapy — Dose escalated Intensity-Modulated Radiation therapy (IMRT) with conventional fractionation, hypofractionation and prostate brachytherapy are allowed.
Drug: Apalutamide — 240 mg PO daily, started the same day as the first LHRHa injection, for 6 months
  Arms: Arm B: ADT + radiation therapy + Apalutamide
Drug: Luteinising Hormone Releasing Hormone analog agonist (LHRHa) — 2 injections of a three-monthly LHRH agonist depot
Drug: Non-steroidal anti-androgen — Non-steroidal anti-androgen (e. g. flutamide, bicalutamide) PO daily for 4 weeks, started 2 weeks before the first LHRH agonist injection
  Arms: Arm A: ADT + radiation therapy

SUMMARY:
The main objective of the trial to determine if the combination of apalutamide with 6 months of androgen deprivation therapy by LHRH agonists in patients with intermediate and limited high-risk, localized prostate cancer receiving primary radiation therapy (RT) results in an improvement of disease-free survival (DFS) evaluated by the treating physician, in comparison to the combination of radiation and androgen deprivation therapy without the addition of apalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma diagnosed by ultrasound guided biopsy of the prostate containing 10-12 cores showing no neuroendocrine component
* Either of: Favorable intermediate risk (according to EAU risk groups): PSA 10-20 ng/mL, -or Gleason score 7 (3 +4) (ISUP Grade 2), or cT2b. Infavorable intermediate risk (according to EAU risk groups): PSA 10-20 ng/mL, -or Gleason score 7 (4+3) (ISUP Grade 3), or cT2b. Limited high risk : PSA > 20 ng/mL or Gleason score >7 (ISUP Grade 4/5)
* M0 by standard imaging work-up
* Scheduled to be treated with primary prostate RT
* WHO Performance Status ≤ 2
* No risk of urinary retention based on the International Prostate Symptom Score (IPSS) : IPSS < 20
* Adequate liver function determined by the following: aspartate aminotransferase (AST), alanine aminotransferase (ALT), < 2.5 x upper limit of normal (ULN). Total bilirubin <1.5 x upper limit of normal (ULN)
* Adequate renal function: creatinine level < 2 x ULN
* Serum albumin ≥ 3.0 g/dL
* Serum potassium ≥ 3.5 mmol/L
* Hemoglobin ≥ 10.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count ≥ 100,000 x 109/L independent of transfusion and/or growth factors within 3 months prior to randomization
* Be able to swallow whole study drug tablets

Exclusion Criteria:

* cT2c, T3, T4 or pelvic lymph nodes involvement, as assessed by CT scan or MRI (cN1) or pelvic lymph node dissection (pN1)
* Previous pelvic irradiation or radical prostatectomy.
* Bilateral orchiectomy
* Prior systemic (e.g., chemotherapy) or procedural (e.g., prostatectomy, cryotherapy) treatment for prostate cancer
* Prior treatment with 5-alpha reductase inhibitors for benign prostatic hypertrophy not discontinued 4 weeks prior to randomization
* Prior treatment with any LHRH agonist or antagonist, bicalutamide, flutamide or nilutamide, enzalutamide, abiraterone acetate, orteronel, galeterone, ketoconazole, aminoglutethimide, estrogens, megestrol acetate, and progestational agents for prostate cancer
* Prior treatment with radiopharmaceutical agents (e.g., strontium-89) or immunotherapy for prostate cancer
* Other malignancy except adequately treated basal cell carcinoma of the skin or other malignancy from which the patient has been cured for at least 5 years.
* History of Ulcerative Colitis, Crohn's Disease, Ataxia Telangiectasia, systemic lupus erythematosus or Fanconi anemia
* History of seizure or condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness ≤ 1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
* Medications known to lower the seizure thresholdmust be discontinued or substituted at least 4 weeks prior to study entry
* Certain risk factors for abnormal heart rhythms/QT prolongation: torsade de pointes ventricular arrhythmias (e.g., heart failure, hypokalemia, or a family history of a long QT syndrome), a QT or corrected QT (QTc) interval > 450 ms at baseline
* Uncontrolled hypertension (systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg); patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Bilateral hip prostheses
* Prior treatment with systemic glucocorticoids ≤ 4 weeks prior to randomization or is expected to require long-term use of corticosteroids during the study
* Use of any investigational agent ≤ 4 weeks prior to randomization
* Current chronic use of opioid analgesics for ≥3 weeks for oral or ≥ 7 days for non-oral formulations
* Major surgery ≤ 4 weeks prior to randomization
* Known or suspected contraindications or hypersensitivity to apalutamide, bicalutamide or LHRHa agonists or any of the components of the formulations
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-10 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 7.8 years from First Patient In (FPI)
  Events for this endpoint include loco-regional recurrence, distant metastases (radiologically or pathologically confirmed), death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Progression-free survival | 7.8 years from First Patient In (FPI)
  includes first events of biochemical failure by Phoenix criteria in addition to the events listed in the primary endpoint DFS
Distant Metastasis-free survival | 7.8 years from First Patient In (FPI)
Overall survival | 7.8 years from First Patient In (FPI)
Prostate cancer specific survival | 7.8 years from First Patient In (FPI)
Prostate-Specific Antigen (PSA) value | 5.5 years from First Patient In (FPI)
  Prostate-Specific Antigen (PSA) value will be assessed at the end of the treatment of each patient
Adverse events graded according to the National Cancer Institute Common Occurrence of Adverse Events | 7.8 years from First Patient In (FPI)
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 4.0
Health-related quality of life | 7.8 years from First Patient In (FPI)
  Health-related quality of life will be evaluated using self-administered EORTC QLQ-C30 questionnaire
Health-related quality of life | 7.8 years from First Patient In (FPI)
  Health-related quality of life will be evaluated using EORTC QLQ-PR25 instruments
Prostate-Specific Antigen (PSA) nadir | 5.5 years from First Patient In (FPI)
  Prostate-Specific Antigen (PSA) nadir will be assessed as the lowest value achievement on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Crehange, Principal Investigator — Centre Georges Francois Leclerc; Michel Bolla, Principal Investigator — CHU de Grenoble - La Tronche - Hôpital A. Michallon, France